CLINICAL TRIAL: NCT02575716
Title: Comparison of Intubating Condition of the Mcgrath Videolaryngoscope With and Without Muscle Relaxant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Piyaporn Vasinanukorn, Dr., Prince of Songkla University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: PSU-561330812
Record Dates: First submitted 2015-10-07; First posted 2015-10-15 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Muscle Relaxant
Keywords: McGrath®; Videolaryngoscope; intubating condition; muscle relaxant; intubation
MeSH Terms: conditions — Muscle Hypotonia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Muscle relaxant (Experimental): Intubation with McGrath video laryngoscope after fentanyl 1.5 mcg/kg, xylocaine 1.5 mg/kg and propofol 3 mg/kg muscle relaxant use rocuronium 0.6 mg/kg
  Interventions: Device: Videolaryngoscope
- Placebo (Placebo Comparator): Intubation with McGrath video laryngoscope after fentanyl 1.5 mcg/kg, xylocaine 1.5 mg/kg and propofol 3 mg/kg placebo use NSS 0.6 mg/kg
  Interventions: Device: Videolaryngoscope

INTERVENTIONS:
Device: Videolaryngoscope — Intubation with McGrath video laryngoscope after muscle relaxant

SUMMARY:
The objective of this study was to evaluate intubating condition using the McGrath® VL Series 5, with and without muscle relaxant

DETAILED DESCRIPTION:
Thirty-four patients with ASA classification I-II, who required oroendotracheal tube intubation, were studied in this prospective, double-blinded, randomized, clinical trial. Anesthesia was induced using fentanyl 1.5 mcg/kg, xylocaine 1.5 mg/kg and propofol 3 mg/kg. Patients were randomly assigned to one of the two groups to receive either rocuronium 0.6 mg/kg or saline intravenously. The Mcgrath® VL intubation was initiated after 90s, when the patients were fully relaxed. The primary outcome was to compare tracheal intubating conditions between two groups. The secondary outcomes were the success rate in the first attempt intubation, time to intubation, the required propofol dose for intubation and anesthetic complications. Statistical analyses were performed using the R program version 2.14.2. The level of statistical significance was set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old.
* ASA class I-II.
* Elective surgery required general anesthesia with oroendotracheal intubation

Exclusion Criteria:

* Suspected or known difficult airway.
* Patient with risk of aspiration with required of rapid sequence induction .
* Plan remained intubation.
* Allergic to drugs used in the study.
* Renal or hepatic disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Intubating condition. | one year
  number of participants with 34 people

SECONDARY OUTCOMES:
Success rate in the first attempt intubation. | one year
Time to intubation | One year
The required propofol dose for intubation without muscle relaxant. | one year
Events during the intubation attempts occurred. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Piyaporn Vasinanukorn, MD., Study Chair — Prince of Songklanagarind University
Locations (1):
- Department of anesthesiology, Hat Yai, Changwat Songkhla, Thailand